CLINICAL TRIAL: NCT05292092
Title: Essential Pro Post-Market Clinical Follow-up Study
Brief Title: Essential Pro PMCF Study ( rEPIC04E )
Acronym: rEPIC04E
Status: Completed | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: Essential Pro PMCF Study
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease (CAD); Ischemic Heart Disease
Keywords: MDR (Medical Device Regulations); PMCF (Post-Market Clinical Follow-up); Paclitaxel eluting coronary balloon dilatation catheter
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Artery Disease (CAD)
  Interventions: Drug: Essential pro

INTERVENTIONS:
Drug: Essential pro — Patients in whom treatment with (Essential Pro) has been attempted

SUMMARY:
Multicenter, prospective, non-randomized, post-market clinical follow-up (PMCF) study to confirm and support the clinical safety and performance of Essential Pro to meet EU Medical Device regulation (MDR) requirements in all the CONSECUTIVE patients treated with Essential Pro.

DETAILED DESCRIPTION:
The objective of this multicenter, prospective, non-randomized, post-market clinical follow-up (PMCF) study is to confirm and support the clinical safety and performance of the Essential Pro in a NON-SELECTED, Real World population under daily clinical practice when used as intended by the manufacturer to meet EU Medical Device regulation requirements for post-market clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated with Essential Pro according to routine hospital practice and following instructions for use
* Informed consent signed

Exclusion Criteria:

• Not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with Essential Pro according to routine hospital practice and following instructions for use
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2025-12-29 (Actual); Study Completion 2026-01-18 (Actual)

PRIMARY OUTCOMES:
Safety Endpoint. Freedom from Target Lesion Failure | 12 months
  Freedom from TARGET LESION FAILURE (TLF), composite endpoint of cardiac death, myocardial infarction (MI) and a new Target Lesion Revascularization (TLR).

SECONDARY OUTCOMES:
Efficacy Endpoint. Freedom from Target Lesion Failure (TLF) | 12 months
  Freedom from TARGET LESION FAILURE (TLF), composite endpoint of Cardiac death, Myocardial infarction, and new Target Lesion Revascularization (TLR).
Freedom from Balloon rupture | During percutaneous coronary intervention (PCI)
  Freedom from Balloon rupture
Freedom from Hypotube rupture | During PCI
  Freedom from Hypotube rupture
Freedom from Complicated withdrawal | During PCI
  Freedom from Complicated withdrawal
Freedom from Coronary perforation | During PCI
  Freedom from Coronary perforation
Freedom from Coronary dissection >C | During PCI
  Freedom from Coronary dissection >C
Freedom from No reflow | During PCI
  Freedom from No reflow
Freedom from Coronary thrombosis | During PCI
  Freedom from Coronary thrombosis

CONTACTS AND LOCATIONS:
Locations (7):
- Spain (7):
  - Hospital Punta de Europa, Algeciras
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de Jerez de la Frontera, Jerez de la Frontera
  - Hospital Universitario de Leon, León
  - Hospital Universitario Regional de Malaga, Málaga
  - Hospital Universitario de Puerto Real, Puerto Real
  - Hospital Universitario Marques de Valdecilla, Santander

REFERENCES:
- [Background] Gruntzig A. Transluminal dilatation of coronary-artery stenosis. Lancet. 1978 Feb 4;1(8058):263. doi: 10.1016/s0140-6736(78)90500-7. No abstract available. PMID 74678
- [Background] Jeger RV, Farah A, Ohlow MA, Mangner N, Mobius-Winkler S, Leibundgut G, Weilenmann D, Wohrle J, Richter S, Schreiber M, Mahfoud F, Linke A, Stephan FP, Mueller C, Rickenbacher P, Coslovsky M, Gilgen N, Osswald S, Kaiser C, Scheller B; BASKET-SMALL 2 Investigators. Drug-coated balloons for small coronary artery disease (BASKET-SMALL 2): an open-label randomised non-inferiority trial. Lancet. 2018 Sep 8;392(10150):849-856. doi: 10.1016/S0140-6736(18)31719-7. Epub 2018 Aug 28. PMID 30170854
- [Background] Wu X, Li L, He L. Drug-Coated Balloon versus Drug-Eluting Stent in Patients with Small-Vessel Coronary Artery Disease: A Meta-Analysis of Randomized Controlled Trials. Cardiol Res Pract. 2021 Apr 13;2021:1647635. doi: 10.1155/2021/1647635. eCollection 2021. PMID 33953973